CLINICAL TRIAL: NCT06620224
Title: Exploring the Impact of Virtual Reality-based Traditional Chinese Acupuncture Treatment on Patient Experience and Doctor-patient Interaction.
Brief Title: Exploring the Impact of VR-based Acupuncture Treatment on Patient Experience and Doctor-patient Interaction.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CMUH113-REC1-147
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Acupuncture; Virtual Reality
Keywords: Traditional Chinese Medicine Acupuncture; Virtual Reality; Technology Acceptance Model; Doctor-Patient Interaction; Medical Quality

STUDY DESIGN:
Intervention Model Description: a non-randomized real world data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant wear the Virtual Reality system (Experimental): Establish a virtual reality acupuncture system, and introduce the technology acceptance model to systematically explore the effectiveness of acupuncture treatment and its related impact on the patient experience and doctor-patient interaction,
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — we only use single group in this study, before the acupuncture treatment, let the participant wear the virtual reality to realize the course of the acupuncture treatment

SUMMARY:
Develop and establish a virtual reality acupuncture system, and introduce the technology acceptance model to systematically explore the impact of acupuncture treatment effectiveness and its related medical experience and doctor-patient interaction

DETAILED DESCRIPTION:
Whether it's Western medicine's surgical treatment or traditional Chinese medicine's acupuncture and acupotomy treatment, for patients preparing to undergo invasive treatment, pre-treatment explanations can improve patient compliance and reduce patient anxiety about disease treatment. The application of virtual reality systems in the medical field is mostly in preoperative training and medical education, while in the field of traditional Chinese medicine, it focuses on acupuncture teaching, with less evaluation of explanations before acupuncture treatment. Therefore, this study will develop and establish a virtual reality acupuncture system, and introduce the technology acceptance model to systematically explore the impact of acupuncture treatment effectiveness and its related medical experience and doctor-patient interaction

ELIGIBILITY:
Inclusion Criteria:

* general public and people see a doctor in the department of acupuncture

Exclusion Criteria:

* participant refusing the intervention of the virtual reality

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Technology Acceptance Model | Immediately
  Measured by the 5-point likert scale:very agree(5), agree(4), neither agree nor disagree(3), disagree(2), very disagree(1)